CLINICAL TRIAL: NCT05024526
Title: Protective Effects of Edaravone Dexborneol in Patients With Acute Ischemic Stroke by Improving Ischemic Penumbra and Collateral Circulation of Hypoperfusion Areas
Brief Title: Protective Effects of Edaravone Dexborneol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lili Cao (Other)
Responsible Party: Sponsor-Investigator, Lili Cao, Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FYQ2021
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Acute Ischemic Stroke
Keywords: edaravone dexborneol; ischemic penumbra; NIHSS; mRS
MeSH Terms: conditions — Ischemic Stroke | interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- edaravone dexborneol group (Experimental)
  Interventions: Drug: edaravone dexborneol or edaravone
- edaravone group (Active Comparator)
  Interventions: Drug: edaravone dexborneol or edaravone

INTERVENTIONS:
Drug: edaravone dexborneol or edaravone — Edaravone dexborneol or edaravone is going to be used in two different groups to compare the efficacy.

SUMMARY:
The patients of acute ischemic stroke were divided into two groups, edaravone dexborneol treatment group and edaravone treatment group. The purpose of this study was to observe the changes of imaging and the improvement of NIHSS and mRS in different groups.

DETAILED DESCRIPTION:
A total of 80 patients with acute ischemic stroke of middle cerebral artery were randomly divided into two groups, edaravone dexborneol treatment group and edaravone treatment group. The mismatch area between the low perfusion area of MRI 3D-ASL and the infarct area of DWI was defined as the ischemic penumbra, and the CBF perfusion pseudo color images with PLD of 1.5s and 2.5s were recorded. The above two CBF perfusion images were subtracted, and the residual area was quantitatively analyzed to reflect the establishment of collateral circulation. We aimed to observe whether there were differences in the improvement of ischemic penumbra and the establishment of collateral circulation between two groups after treatment. Besides, the improvment of NIHSS and mRS was also observed in different periods.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 50 to 80 years old;
2. Patients diagnosed as acute ischemic stroke according to Chinese guidelines for the diagnosis and treatment of acute ischemic stroke 2018 and who met the requirements of middle cerebral artery blood supply area infarction (except deep perforator disease) without treatment;
3. Brain MR showed that the low perfusion area of ASL was at least 20% larger than that of DWI core infarct area, and the contralateral mirror brain tissue was basically normal;
4. NIHSS score was between 4 to 24;
5. Patient or their legal representatives were willing to sign the informed consent form.

Exclusion Criteria:

1. Serious mental abnormality, complicated with heart, lung, liver, renal insufficiency or malignant tumor and other serious diseases;
2. Combined with cerebral vascular malformation or cerebral hemorrhage;
3. Pregnant or lactating women;
4. Allergic to edaravone or dexborneol;
5. There are interactions between the drugs being taken by patients and the study drug or affect the clinical trial parameters.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
image changes in different groups | 7 days

SECONDARY OUTCOMES:
NIHSS changes in different groups | 7days，14 days, 90 days
mRS changes in different groups | 7days，14 days, 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Qing Fang, MD, Principal Investigator — Shandong Provincial Qianfoshan Hospital，The First Affiliated Hospital of Shandong First Medical University
Locations (1):
- Shandong Provincial Qianfoshan Hospital，The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No